CLINICAL TRIAL: NCT03905005
Title: Jaw Reconstruction With Printed Titanium and Free Tissue Transfer
Acronym: JaW PrinT
Status: Completed | Type: Observational
Sponsor: University of South Wales (Other)
Responsible Party: Sponsor
Other Study IDs: 241919; 38098 (Other: CPMS (UK central portfolio management system))
Record Dates: First submitted 2019-03-29; First posted 2019-04-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Neoplasm, Oral; Osteoradionecrosis of Jaw; Mandibular Diseases; Jaw Cancer; Jaw Diseases; Surgery
MeSH Terms: conditions — Mouth Neoplasms; Mandibular Diseases; Jaw Neoplasms; Jaw Diseases | interventions — Mandibular Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-flexed reconstruction plate: Patients who undergo mandibular reconstruction using a pre-flexed osseosynthesis reconstruction plate along with free-tissue transfer for reconstruction of a mandibular continuity defect.
  Interventions: Procedure: Mandibular reconstruction with free tissue transfer.
- Printed reconstruction plate: Patients who undergo mandibular reconstruction using a 3D-printed reconstruction plate made by selective laser melting (SLM), along with free-tissue transfer for reconstruction of a mandibular continuity defect.
  Interventions: Procedure: Mandibular reconstruction with free tissue transfer.

INTERVENTIONS:
Procedure: Mandibular reconstruction with free tissue transfer. — Mandibular reconstruction with free tissue transfer (free-flap bony reconstruction) requires the use of a titanium plate to secure bony segments until bony healing is complete. Plates are made of titanium but can be customised to the anatomical shape of the mandible by two different techniques: flexing (bending) of the plate before surgery, or printing of the plate from titanium alloy powder bed fusion techniques (additive manufacturing, such as selective laser melting).

SUMMARY:
JaW PrinT is a prospective observational cohort study evaluating the effectiveness of two different techniques of mandibular reconstruction.

DETAILED DESCRIPTION:
JaW PrinT is a 'real-world' prospective observational pilot study, evaluating the clinical effectiveness, usability and economics of two approaches to mandibular reconstruction surgery (using flexed titanium versus printed titanium patient-specific osseosynthesis plates). Patient participants will be recruited prospectively over a minimum period of 18 months (with observation of at least 10 participants in each treatment pathway). The figures are based upon the historical clinical practice of the research site, with both techniques in equal use; choice depending on resources, surgical training requirements and surgeon's clinical preference.

As a purely observational study, treatment choice will be made in the normal clinical manner and will in no way be influenced by the study itself.

Participants will be followed up at their routine outpatient clinics (6 weeks, 6 months and 1 year postoperatively) with prospective outcomes data collection.

Participants will be recruited prospectively as they present as new patient cases to the Maxillofacial and Head & Neck cancer multidisciplinary team (MDT) clinics. Once a potential patient participant has been given his/her diagnosis and it is confirmed by the principal investigator (PI) that he/she meets the inclusion criteria, clinic staff will provide the potential participant with an invitation letter introducing the study as well as a patient information sheet and consent form (explaining the available options of participating or refraining from the study). Patients will be allowed up to 24 hours to decide whether or not to participate as to avoid any impact/delay on the scheduling of their clinical treatment. The PI will obtain written informed consent from willing participants.

Upon recruitment, provision of informed consent and collection of baseline data, as per standard clinical practice, the patient participant's CT scan data is used to produce a virtual surgical plan for the mandibular resection and fibular free-flap reconstruction. Once the clinically optimal reconstructive surgical plan is established by the surgeon and technician, the choice of surgical approach will be made in the routine clinical manner by the surgeon: Pathway A (pre-flexed customized mandibular reconstruction plate and cutting guides) or to pathway B (SLM customized mandibular reconstruction plate and cutting guides). Both treatment pathways are already part of routine/standard clinical practice at the research site.

The expected/planned patient numbers for this study are based upon the historical workload of the department, typically at 10-20 cases annually. A recruitment period of 18 months with follow-up for 1 year fits within the time constraints of the postgraduate student investigator's PhD timeline.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Able to provide informed consent
* A planned fibular free-flap reconstruction of the mandible
* Planned post operative surveillance CT scan 6 months following surgery

Exclusion Criteria:

* Clinically unfit or inappropriate (based upon prognosis/life expectancy) for reconstruction using free tissue transfer techniques
* Patients with planned surgical defects involving formal reconstruction of the condyle. (Clinical use of printed plates for condylar reconstructions would in effect be 'off-licence' and non-standard treatment which is beyond the remit of an observational research study).
* Flap failure within the study follow-up period, as this would require early removal of the flap and therefore preclude collection of follow-up outcome data. However, any flap failures (and associated clinical complications/events) will be recorded and reported.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the study site region requiring free-flap reconstruction of the mandible (e.g. for tumour or osteoradionecrosis):
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Dimensional accuracy | 6 months
  Dimensional accuracy of the bony reconstruction, as demonstrated by comparing 6 months postoperative CT scan DICOM data with a presurgical digital surgical plan.

SECONDARY OUTCOMES:
Duration of surgery | 1 day (day of surgery)
  The impact of surgical technique (pathway A or B) on the duration of insetting the bony flap into the mandibular continuity defect.
Operator's rating of usability/confidence/satisfaction with technique | 1 day (day of surgery)
  Using 5 point Likert scale ratings of ease of flap preparation, ease of locating the reconstruction plate on the fibula, confidence with technique, ease of mandibular reconstruction, ease of locating the reconstruction plate on the mandible, bony apposition of fibula-fibula and fibula-mandible osteotomies as planned, satisfaction with morphology of reconstructed mandible, confidence with technique overall (strongly disagree, disagree, neither agree nor disagree, agree, strongly agree).
Need to make adjustments to reconstructive surgical plan intraoperatively | 1 day (day of surgery)
  List of all required adjustments to the planned reconstructive surgical procedure (e.g. trimming of osteotomies etc.) are recorded.
Complications | 1 year postoperatively
  Incidence of intra/peri/post-operative complications are recorded (e.g. infection, plate exposure, prolonged hospital stay, non-union etc.)
Qualitative evaluation of dental occlusal relationship and feasibility of dental implant rehabilitation | 1 year postoperatively
  Qualitative Evaluation of changes in dental occlusion by evaluating dental plaster of Paris models (presence or absence of "malocclusion" pre and post-operatively) PLUS assessment/rating of feasibility of dental implant rehabilitation in relation to actual bony reconstruction using a 5 point likert scale (strongly disagree, disagree, neither agree nor disagree, agree, strongly agree)
Patient reported quality of life relating to appearance | Baseline, 6 weeks, 6 months, 1 year postoperatively
  Subjective scoring of patient's own perceptions of their quality of life relating to their appearance using the Derriford Appearance Scale
Patient perceived quality of life relating to mood | Baseline, 6 weeks, 6 months, 1 year postoperatively
  University of Washington v4.0 questionnaire score.
Financial implications of surgical technique | Separately for duration of inpatient hospital stay (typically 2 weeks) and for the total 1 year study follow-up period (from identification of participant to completion of patient's participation).
  Evaluation of cost differences (if any) between patient groups
Patient perceived quality of life relating to oral function | Baseline, 6 weeks, 6 months, 1 year postoperatively
  Liverpool oral rehabilitation questionnaire scores.
objective quantitative evaluation of facial symmetry | Baseline, 6 weeks, 6 months, 1 year postoperatively
  stereophotogrammetry to assess facial symmetry.

CONTACTS AND LOCATIONS:
Overall Officials: M Williams, PhD, Study Chair — University of South Wales; A Goodson, MBBS, Study Director — University of South Wales; M Kittur, MBBS, Principal Investigator — Morriston Hospital, ABMU Health Board
Locations (1):
- Morriston Hospital, Swansea, United Kingdom

DOCUMENTS (1):
  • Study Protocol (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT03905005/Prot_000.pdf